CLINICAL TRIAL: NCT03092830
Title: Molecular Characterization of Cutaneous Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0515-15-RMC
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Squamous Cell Carcinoma; Basal Cell Carcinoma
Keywords: SCC; BCC; DNA; RNA; HEDGE HOG; epidermal growth factor receptor
MeSH Terms: conditions — Carcinoma, Squamous Cell; Carcinoma, Basal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA or RNA which will be produced from skin biopsy specimens of SCC,BCC
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1-arm, 500 participates: Molecular testing of DNA/RNA from skin tumors, SCC/BCC
  Interventions: Genetic: Molecular testing of DNA/RNA from skin tumors, SCC/BCC

INTERVENTIONS:
Genetic: Molecular testing of DNA/RNA from skin tumors, SCC/BCC — Molecular testing of DNA/RNA from skin tumors, SCC/BCC

SUMMARY:
The objective is to find genes which are responsible for the appearance of skin tumors (sCC, BCC) and it will be the basis for prediction of the disease and response to the treatment

DETAILED DESCRIPTION:
Prospective, 1-arm, 500 participates above 18 age with skin tumor affliction sCC and BCC type.

ELIGIBILITY:
Inclusion Criteria:

* patient that have sCC and BCC tumors
* above 18 years old

Exclusion Criteria:

* below 18 years old
* pregnant women
* children or person without judgment ability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: above 18 years old with Scc and BCC skin tumors not pregnant women and no children or any person without judgment ability
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-03-29 (Actual); Primary Completion 2020-08-07 (Estimated); Study Completion 2020-08-07 (Estimated)

PRIMARY OUTCOMES:
Molecular Characterization of cutaneous tumors | 5 years
  samples from subjects

CONTACTS AND LOCATIONS:
Overall Officials: DR Dean Ad EL, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- RabinMC, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Winder M, Viros A. Mechanisms of Drug Resistance in Melanoma. Handb Exp Pharmacol. 2018;249:91-108. doi: 10.1007/164_2017_17. PMID 28275910